CLINICAL TRIAL: NCT04374474
Title: Olfactory Retraining Therapy and Budesonide Nasal Rinse for Anosmia Treatment in Patients Post-CoVID 19. A Randomized Controlled Trial
Brief Title: Anosmia Rehabilitation in Patients Post Coronavirus Disease (COVID 19)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn before any enrollment (site's research goals adjustments).
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anosmia_CoVID 19
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-10

CONDITIONS: Olfactory Disorder
Keywords: anosmia; hyposmia; CoVID19; post-viral anosmia; snap and sniff olfactory test; budesonide
MeSH Terms: conditions — Anosmia; COVID-19 | interventions — Olfactory Training; Nasal Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Sham Comparator): The participants, randomly assigned to this arm, will receive a paper hand-out about post-viral anosmia with instructions to smell common household items (current care). Besides, it will be prescribed nasal irrigation twice a day.
  Interventions: Other: smell household Items; Other: Nasal Irrigation
- Olfactory Retraining Group (Experimental): The participants, randomly assigned to this arm, will receive instructions on olfactory retraining and will also be given an essential oil retraining kit, which they will use twice a day. Besides, it will be prescribed nasal irrigation twice a day.
  Interventions: Other: Olfactory retraining; Other: Nasal Irrigation
- Olfactory Retraining_Budesonide Group (Experimental): The participants, randomly assigned to this arm, will receive instructions on olfactory retraining, the olfactory training kit and it will be prescribed nasal irrigation with Budesonise, twice a day.
  Interventions: Other: Olfactory retraining; Drug: corticosteroid nasal irrigation

INTERVENTIONS:
Other: Olfactory retraining — Olfactory retraining Olfactory training is performed by exposing patients twice daily to essential oils with four specific odors, present in glass jars with soaked cotton pads: phenyl ethyl alcohol, rose; eucalyptol, eucalyptus; citronellal, lemon; eugenol, cloves.
  Other Names: essential oils kit; smell training
  Arms: Olfactory Retraining Group; Olfactory Retraining_Budesonide Group
Drug: corticosteroid nasal irrigation — Nasal irrigation with corticosteroid (budesonide) consists of 240-mL nasal irrigation with Pulmicort Respules (0.5mg) across both nose sides via NeilMed Sinus Rinse bottle (Santa Rosa, California, USA).
  Other Names: Budesonide nasal irrigation
  Arms: Olfactory Retraining_Budesonide Group
Other: smell household Items — Participants will receive a paper hand-out about post-viral anosmia with instructions to smell common household items
  Arms: Control Group
Other: Nasal Irrigation — Participants from all three groups will use nasal rinse (NeilMed Sinus Rinse) two times a day.
  Other Names: Nasal Rinse
  Arms: Control Group; Olfactory Retraining Group

SUMMARY:
The study will be a randomized controlled trial, involving patients with hyposmia/anosmia of onset immediately after an upper respiratory viral illness, assigned to three distinct study arms. Nasal irrigations will be prescribed to all three groups (BID). In addition, one arm will receive a paper hand-out about post-viral anosmia with instructions to smell common household items (current care) and act as a control group. The second group will receive an essential oil retraining kit, whereas the third group will receive the same olfactory training kit and a prescription to use budesonide with the nasal irrigations. Olfactory scores will be tested at the enrollment, 3 months and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Hyposmia/anosmia of onset immediately after an upper respiratory viral illness confirmed on Snap n' Sniff threshold testing,
* Capable, in the opinion of the primary investigator, of providing informed consent to participate in the study. Participants are required to sign an informed consent form indicating they understand the purpose and nature of the study, and that they are willing to participate.

Exclusion Criteria:

* active cigarette smoker
* chronic rhinosinusitis
* head trauma with loss of consciousness
* inability to read/understand English
* previous hyposmia/anosmia complaint
* pregnancy
* previous sinus
* skull base or brain surgery
* current participation in another clinical trial at the time of initial visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-10 (Estimated); Primary Completion 2021-12-10 (Estimated); Study Completion 2022-03-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Snap and Sniff Threshold Test at 3 months | 3 months
  Score from the Snap and Sniff Olfactory Test results
Change from baseline Smell Identification Test (SIT) at 3 months | 3 months
  Score from the Smell Identification test results.
Change from Baseline Snap and Sniff Threshold Test at 6 months | 6 months
  Score from the Snap and Sniff Olfactory Test results
Change from baseline Smell Identification Test (SIT) at 6 months | 6 months
  Score from the Smell Identification test results.

SECONDARY OUTCOMES:
Change from baseline QOD-NS at 3 months | 3 months
  Scores from the short version of the Questionnaire of Olfactory Disorders Negative Statements (QOD-NS)
Change from baseline SF-36 health survey at 3 months | 3 months
  Short Form 36 Health Survey scores
Change from baseline QOD-NS at 6 months | 6 months
  Scores from the short version of the Questionnaire of Olfactory Disorders Negative Statements (QOD-NS)
Change from baseline SF-36 health survey at 6 months | 6 months
  Short Form 36 Health Survey scores
Adherence to the Study Protocol | 6 months
  Adherence comparison between participants post-CoVID 19 and patients post other viral infections.
Recovery | 6 months
  Compare the rate of recovery between post-COVID 19 patients and patients post other viral infections.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Sowerby, MD, FRCSC, Principal Investigator — Western University
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Background] Vennemann MM, Hummel T, Berger K. The association between smoking and smell and taste impairment in the general population. J Neurol. 2008 Aug;255(8):1121-6. doi: 10.1007/s00415-008-0807-9. Epub 2008 Jul 28. PMID 18677645
- [Background] Croy I, Nordin S, Hummel T. Olfactory disorders and quality of life--an updated review. Chem Senses. 2014 Mar;39(3):185-94. doi: 10.1093/chemse/bjt072. Epub 2014 Jan 15. PMID 24429163
- [Background] Konstantinidis I, Tsakiropoulou E, Bekiaridou P, Kazantzidou C, Constantinidis J. Use of olfactory training in post-traumatic and postinfectious olfactory dysfunction. Laryngoscope. 2013 Dec;123(12):E85-90. doi: 10.1002/lary.24390. Epub 2013 Oct 4. PMID 24114690
- [Background] Nguyen TP, Patel ZM. Budesonide irrigation with olfactory training improves outcomes compared with olfactory training alone in patients with olfactory loss. Int Forum Allergy Rhinol. 2018 Sep;8(9):977-981. doi: 10.1002/alr.22140. Epub 2018 Jun 14. PMID 29901865
- [Background] Mattos JL, Edwards C, Schlosser RJ, Hyer M, Mace JC, Smith TL, Soler ZM. A brief version of the questionnaire of olfactory disorders in patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2019 Oct;9(10):1144-1150. doi: 10.1002/alr.22392. Epub 2019 Aug 20. PMID 31430061
- See also: Snap and Sniff threshold test informative website — https://sensonics.com/product/snap-sniff-odor-threshold-test/